CLINICAL TRIAL: NCT01404585
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy, Safety, Tolerability, and Pharmacokinetics of BMS-817399 in Adults With Active, Moderate to Severe Rheumatoid Arthritis and Inadequate Response to Methotrexate
Brief Title: Proof-of-Concept Study With BMS-817399 to Treat Moderate to Severe Rheumatoid Arthritis
Acronym: RA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM126-004; 2011-002024-40 (EudraCT Number)
Record Dates: First submitted 2011-07-27; First posted 2011-07-28 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — 1-(1-(4-(4-chlorophenyl)-4-hydroxy-3,3-dimethylpiperidin-1-yl)-3-methyl-1-oxobutan-2-yl)-3-(2-hydroxy-2-methylpropyl)urea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Arm 2: BMS-817399 (200 mg) (Experimental)
  Interventions: Drug: BMS-817399
- Arm 3: BMS-817399 (400 mg) (Experimental)
  Interventions: Drug: BMS-817399

INTERVENTIONS:
Drug: Placebo — Tablets, Oral, 0 mg, twice daily, 12 weeks
  Arms: Arm 1: Placebo
Drug: BMS-817399 — Tablets, Oral, 200 mg, twice daily, 12 weeks
  Arms: Arm 2: BMS-817399 (200 mg)
Drug: BMS-817399 — Tablets, Oral, 400mg, twice daily, 12 weeks
  Arms: Arm 3: BMS-817399 (400 mg)

SUMMARY:
The purpose of this study is to assess whether BMS-817399 in combination with Methotrexate is effective in treating moderate to severe rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, 18 years of age or older, with rheumatoid arthritis (RA) for at least 6 months prior to screening
* Subjects must have a tender joint count of at least 6 (28 joint count), swollen joint count of at least 6 (28 joint count) at screening. All subjects must have clinical evidence of synovitis in one hand/wrist at screening
* Serum C-reactive protein (hsCRP) above upper limits of normal at screening
* Subjects must have been treated with and tolerated Methotrexate (MTX) therapy at a weekly oral or parenteral dose ≥ 10 mg for ≥ 4 months prior to screening. Dose must be stable, with no change in route of administration, for ≥ 6 weeks prior to randomization. A MTX weekly dose as low as 7.5 mg is permitted if intolerance to doses ≥10 mg has been documented in the subject's medical history
* Subjects must be receiving folic acid, folinic acid, or leucovorin supplementation at a stable dose for at least 4 weeks prior to randomization
* Subjects who were previously treated with up to two tumor necrosis factor α (TNF-α) inhibitors
* If taking antimalarials (e.g. hydroxychloroquine or chloroquine), subject must have been on a stable dose for ≥ 4 months prior to randomization
* If taking non-steroidal anti-inflammatory drugs (NSAIDs), subjects must have been on stable doses for ≥ 2 weeks prior to randomization
* If taking oral corticosteroids, daily doses must be ≤ 10 mg/day of prednisone or equivalent and stable for ≥ 4 weeks before randomization
* Subject is willing to participate to the study and has signed the informed consent prior to undergoing any screening procedures
* Women of childbearing potential (WOCBP) and men must agree to use at least two acceptable methods to avoid pregnancy for the entire study period and until 60 days (for women) and 90 days (for men) after the last dose of BMS-817399. WOCBP must have a negative urine pregnancy test at screening, randomization and at scheduled visits throughout the study

Exclusion Criteria:

* Arthritis onset prior to 16 years of age or subjects with documented juvenile RA
* Subjects who are bed- or wheelchair-bound
* Subjects with other autoimmune diseases or arthritis syndromes
* Women who are pregnant, breastfeeding or with a positive pregnancy test at screening or prior to randomization
* Subjects who have any condition that could impact upon the absorption of study drug (i.e., gastric stapling, duodenal surgery, malabsorption syndrome)
* Subjects with a history of, or a concurrent severe, progressive, or uncontrolled disease (other than RA) that in the opinion of the investigator might place the subject at unacceptable risk for participation in this study
* Subjects who have present or previous (last 5 years) malignancies, except history of cured squamous or basal skin cell carcinoma or cured breast or cervical cancer
* Subjects at risk for tuberculosis (TB) or with evidence of TB clinical history, chest X rays or tuberculin skin test
* Subjects with evidence of active or latent bacterial or viral infections (including human immunodeficiency virus); Positive blood screen for hepatitis B surface antigen or hepatitis C antibody
* Subjects with any serious bacterial infection within the last 2 months, unless treated and resolved with antibiotics
* Subjects who have clinically significant drug or alcohol abuse or known cirrhosis including alcoholic cirrhosis
* If a subject has received any of the following treatments, the indicated washout period prior to randomization must be followed:

  1. Oral or injectable azathioprine, gold, D-Penicillamine, cyclosporine, anakinra, etanercept, parenteral or intra-articular corticosteroids: 30 days
  2. Leflunomide: 6 months unless an active washout with Cholestyramine has been performed
  3. Mycophenolate mofetil, cyclophosphamide, tacrolimus or other immunosuppressant: 3 months
  4. Adalimumab, Infliximab, Golimumab, Certolizumab pegol, Abatacept or Tocilizumab: 60 days
  5. Rituximab or any B-cell depleting agent: 1 year
* Use CYP3A4 inhibitors or inducers during the study
* Subjects with alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 1.5x upper limit of normal (ULN), total bilirubin ≥ 1.4x ULN, estimated glomerular filtration rate (GFR) < 50 mL/min/1.73m2, hemoglobin < 10.0 g/dL, white blood cell count < 3,500/mm3, absolute neutrophil count < 1,700/mm3 or platelets < 125,000/mm3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2011-09; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Disease Activity Score using 28 joint count and C Reactive Protein (DAS28-CRP) change from baseline of BMS-817399 versus placebo | Baseline and at 12 weeks

SECONDARY OUTCOMES:
Safety assessments will be based on adverse event reports and the results of vital sign measurements, electrocardiogram, physical examinations, and clinical laboratory tests | 16 weeks
Proportion of subjects achieving 20% American College of Rheumatology (ACR) response in each treatment group | Day 15
Proportion of subjects achieving 20% ACR response in each treatment group | Day 29
Proportion of subjects achieving 20% ACR response in each treatment group | Day 57
Proportion of subjects achieving 20% ACR response in each treatment group | Day 85
Proportion of subjects achieving 50% ACR response in each treatment group | Day 15
Proportion of subjects achieving 50% ACR response in each treatment group | Day 29
Proportion of subjects achieving 50% ACR response in each treatment group | Day 57
Proportion of subjects achieving 50% ACR response in each treatment group | Day 85
Proportion of subjects achieving 70% ACR response in each treatment group | Day 15
Proportion of subjects achieving 70% ACR response in each treatment group | Day 29
Proportion of subjects achieving 70% ACR response in each treatment group | Day 57
Proportion of subjects achieving 70% ACR response in each treatment group | Day 85
Percent change from baseline in disability index of the Health Assessment Questionnaire (HAQ-DI) | Baseline and Day 15
Percent change from baseline in disability index of the Health Assessment Questionnaire (HAQ-DI) | Baseline and Day 29
Percent change from baseline in disability index of the Health Assessment Questionnaire (HAQ-DI) | Baseline and Day 57
Percent change from baseline in disability index of the Health Assessment Questionnaire (HAQ-DI) | Baseline and Day 85
To assess the minimum observed concentration (Cmin) of BMS-817399 | Day 15, Day 29, Day 57 and Day 85

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (25):
- United States (5):
  - Desert Medical Advances, Palm Desert, California
  - Sarasota Arthritis Research Center, Sarasota, Florida
  - Paramount Medical Research & Consulting, Llc, Middleburg Heights, Ohio
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - Pharma Resource, East Providence, Rhode Island
- Argentina (3):
  - Local Institution, Buenos Aires, Buenos Aires
  - Local Institution, Capital Federal, Buenos Aires
  - Local Institution, San Miguel de Tucumán, Tucumán Province
- Mexico (5):
  - Local Institution, Tijuana, Estado de Baja California
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, D.f., Mexico City
  - Local Institution, San Luis Potosí City, San Luis Potosí
  - Local Institution, Mérida, Yucatán
- Russia (2):
  - Local Institution, Moscow
  - Local Institution, Yaroslavl
- South Africa (4):
  - Local Institution, Pretoria, Gauteng
  - Local Institution, Durban, KwaZulu-Natal
  - Local Institution, Panorama, Western Cape
  - Local Institution, Pinelands, Western Cape
- South Korea (3):
  - Local Institution, Daegu
  - Local Institution, Gwangju
  - Local Institution, Seoul
- Spain (3):
  - Local Institution, Córdoba
  - Local Institution, Santiago de Compostela
  - Local Institution, Seville

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx